CLINICAL TRIAL: NCT00001717
Title: Influences on HIV Infected Subjects' Willingness to Participate in Research and Ability to Give Informed Consent
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980131; 98-CC-0131
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections
Keywords: Compensation; Motivations; Volunteers; HIV
MeSH Terms: conditions — HIV Infections

SUMMARY:
This protocol seeks to better understand the various factors which influence an HIV infected individual's decision to participate in clinical research, and especially how the offer of payment influences the decision to participate and understanding of the risks, benefits and purpose of the research. Subjects will be HIV infected individuals participating in or being screened for participation in intramural HIV studies being conducted by the NIAID, CCMD, and NCI. Willing subjects will be recruited from studies that offer payment and comparable studies that do not pay. The primary methodology is an interview via a survey schedule. Use of the interview schedule will be preceded by a focus group of about 7-10 individuals and pretesting of the survey instrument. Paid and unpaid subjects will be compared with respect to motivations, understanding, willingness to withdraw, and sociodemographics.

DETAILED DESCRIPTION:
This protocol seeks to better understand the various factors which influence an HIV infected individual's decision to participate in clinical research, and especially how the offer of payment influences the decision to participate and understanding of the risks, benefits and purpose of the research. Subjects will be HIV infected individuals participating in or being screened for participation in intramural HIV studies being conducted by the NIAID, CCMD, and NCI. Willing subjects will be recruited from studies that offer payment and comparable studies that do not pay. The primary methodology is an interview via a survey schedule. Use of the interview schedule will be preceded by a focus group of about 7-10 individuals and pretesting of the survey instrument. Paid and unpaid subjects will be compared with respect to motivations, understanding, willingness to withdraw, and sociodemographics.

ELIGIBILITY:
Those HIV seropositive subjects participating in or being screened for participation in selected NIAID or NCI intramural HIV studies will be eligible for participation in this study.

Eligible subjects are those willing and able to provide their own informed consent.

No subjects that are unable to speak English or are unable or unwilling to communicate with investigators for any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225
Dates: Start 1998-07; Study Completion 2000-07

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ayd FJ Jr, Calabresi P. Motivations and rewards for volunteering to be an experimental subject. Clin Pharmacol Ther. 1972 Sep-Oct;13(5):771-81. doi: 10.1002/cpt1972135part2771. No abstract available. PMID 5054323
- [Background] Bigorra J, Banos JE. Weight of financial reward in the decision by medical students and experienced healthy volunteers to participate in clinical trials. Eur J Clin Pharmacol. 1990;38(5):443-6. doi: 10.1007/BF02336681. PMID 2379528
- [Background] Ross MW, Jeffords K, Gold J. Reasons for entry into and understanding of HIV/AIDS clinical trials: a preliminary study. AIDS Care. 1994;6(1):77-82. doi: 10.1080/09540129408258027. PMID 8186281